CLINICAL TRIAL: NCT01736670
Title: An Investigator-Initiated Study to Assess the Cooling Effect of Triamcinolone Acetonide Aerosol When Used for Steroid-Responsive Dermatoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patel, Rita Vikram, M.D. (Individual)
Collaborators: Ranbaxy Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GCO#11-0008
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Acute Steroid Responsive Dermatoses; Chronic Steroid Responsive Dermatoses
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acute Steroid Responsive dermatitis (Experimental): 10 patients with acute steroid-responsive dermatoses
  Interventions: Drug: Triamcinolone Acetonide spray; Drug: Triamcinolone acetonide cream; Drug: Alcohol spray
- Chronic Steroid Responsive Dermatits (Experimental): 10 patients with chronic steroid-responsive dermatoses
  Interventions: Drug: Triamcinolone Acetonide spray; Drug: Triamcinolone acetonide cream; Drug: Alcohol spray
- Control, Otherwise healthy (Active Comparator): 10 healthy controls
  Interventions: Drug: Triamcinolone Acetonide spray; Drug: Triamcinolone acetonide cream; Drug: Alcohol spray

INTERVENTIONS:
Drug: Triamcinolone Acetonide spray
Drug: Triamcinolone acetonide cream
Drug: Alcohol spray

SUMMARY:
Triamcinolone acetonide is a mid-potency, class 4/5 topical corticosteroid that is available in a spray formulation (Triamcinolone Acetonide Spray, T Spray). It is indicated for the relief of inflammatory and pruritic manifestations of corticosteroid-responsive dermatoses. Unlike more potent steroid products, T Spray has no time limitations on its use; therefore, it is commonly used to treat flares in psoriasis, atopic dermatitis, seborrheic dermatitis, and contact dermatitis.

In contrast to creams and ointments, T Spray can easily cover large and hard-to-reach areas of the body. Its optional nozzle directs application of the medication to precise areas without affecting nearby areas. Patients requiring a mid-potency corticosteroid for lesions on the scalp, back, intertriginous folds, large areas, or areas that require precise application would benefit from the T Spray formulation. In the time since the introduction of T Spray to dermatology, other topical corticosteroids have entered the market, but T Spray remains the only mid-potency corticosteroid available in a spray formulation.

In a recently published open-label, non-comparator study involving 42 patients with chronic steroid-responsive dermatoses, T Spray was used up to four times a day for 28 days. Improvement of lesions after one week of treatment was experienced by 85% of patients, and 95% of subjects preferred the spray over creams and ointment. Most importantly, 56% of patients reported an anti-pruritic cooling effect which was experienced upon application.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years old and in good general health, as confirmed by a medical history
2. A clear diagnosis of the chronic steroid-responsive dermatosis (i.e. psoriasis, atopic dermatitis) or acute steroid-responsive dermatosis (i.e. contact dermatitis, first-degree burn) must have been previously established and patients must have a target lesion that can be assessed for severity of inflammation
3. Females of childbearing potential must have a negative urine pregnancy test to participate in the study
4. Subjects must be able to understand the requirements of the study and sign an informed consent prior to study procedures

Exclusion Criteria:

1. Subjects who are pregnant and/or nursing
2. Subjects with a known hypersensitivity to any component of the T Spray
3. Subjects who are using any medication or have a disease which in the judgment of the investigator will interfere with the conduct or interpretation of the study
4. Subjects with any of the following pathologies: cold urticaria, cryoglobulinemia, Raynaud's phenomena, or Paroxysmal cold hemoglobulinuria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Skin Surface Temperature Change | 1 month
  By using an infrared video camera, to assess whether Triamcinolone Acetonide Spray's (T Spray) reduces in skin surface temperature (SST) when applied as indicated, for a two-second spray interval, to either acute or chronic steroid-responsive dermatoses

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States